CLINICAL TRIAL: NCT06943209
Title: Assessing the faiSAbility of a Peer-to-peer Contraceptive Education Program on Social Networks Aimed at 15- to 19-year-old High School Students in GuAdeloupe and La RéunIon: a Before-after SAPLAI Pilot Study
Brief Title: SAPLAI : Assessing the faiSAbility of a Peer-to-peer Contraceptive Education Program on Social Networks Aimed at 15- to 19-year-old High School Students in GuAdeloupe and La RéunIon
Acronym: SAPLAI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/CHU/05; 2025-A00358-41 (Other: ID-RCB)
Record Dates: First submitted 2025-04-14; First posted 2025-04-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Contraception Behavior
Keywords: influencers; peer educators; students; sexual health
MeSH Terms: conditions — Contraception Behavior | interventions — Early Intervention, Educational; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Influencer peer group: Creation of a contraception education program and posting of messages/videos on social networks
  Interventions: Other: Creation of a contraception education program and post on social networks for high school students; Other: Survey and questionnaires
- All high school students: All high school students in the 4 selected classes
  Interventions: Other: Education program; Other: Survey and questionnaires

INTERVENTIONS:
Other: Creation of a contraception education program and post on social networks for high school students — Training of peer influencers and program design.
  Groups: Influencer peer group
Other: Education program — View videos/messages created by peer influencers on social networks
  Groups: All high school students
Other: Survey and questionnaires — Respond to the sexual health and contraception knowledge survey and the education program satisfaction survey

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of a contraception education program delivered by peers via social networks to high school students.

Our primary hypothesis is that the implementation of a peer-led contraceptive education program via social networks is a feasible approach in high schools on Reunion Island and Guadeloupe, as part of a before-and-after study.

Our secondary hypotheses concern the evaluation of adoption, exploratory efficacy (on knowledge, attitudes and practices), acceptability and fidelity of the peer-led education program via social networks among high school students in La Réunion and Guadeloupe.

Participants will :

* Participate in a focus group to explore their views and experiences regarding the value of a peer educator as a source of sexual and reproductive health information.
* answer questionnaires on their knowledge of sexual health
* A selected group (peer influencers): Create educational content (after a training period) on sexual health, and particularly contraception, to be broadcast on social networks.
* Take note of the program distributed on the networks by the peer influencers (for 3 months)
* Fill in questionnaires on their knowledge of sexual health, after the program.

ELIGIBILITY:
Inclusion Criteria:

* HIGH SCHOOL STUDENTS
* Young men and women aged between 15 and 19
* Living in La Réunion or Guadeloupe
* Enrolled in one of the selected vocational high schools and whose school principal agrees to take part in the program
* Who have agreed to take part in the study
* Who have received written consent from a parent or guardian.

PEER INFLUENCERS

* Young men and women aged between 15 and 19
* Living in La Réunion or Guadeloupe
* Enrolled in one of the selected vocational high schools and whose school principal agrees to participate in the program
* Selected in seconde class and admitted to première class
* Have been chosen as a peer
* Have a sense of self-efficacy in the use of computers
* Have good communication skills
* Possession of a video-capable smartphone
* Having agreed to take part in the study
* Written consent from a parent or guardian

Exclusion Criteria:

- Involved in other similar programs

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: High school students aged 15 to 19 from 4 selected classes (2 in Rénuon and 2 in Guadeloupe)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the contraceptive education program, measured by the commitment rate of peer influencers. | From date of enrollment until the end of the programm and its evaluation, assessed up to 15 months
  This rate corresponds to the percentage of tasks completed out of the total planned tasks to be carried out by peers in the contraception education program over 3 months. We consider that the program will be feasible if at least 70% of the tasks planned by the peer educators are completed during the 3 months of intervention with high school students.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle REYNAUD, Principal Investigator — CHU REUNION
Locations (2):
- LYCEE POLYVALENT- NORD GRANDE TERRE de PORT-LOUIS, Port-Louis, Guadeloupe, Guadeloupe
- Vue Belle vocational school,, Saint-Paul, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynaud D, Lenclume V, Bertrand L, Balaga AM, Laboureur E, Bruneau L. Feasibility of a peer-led educative programme on contraception using social media for high school students: a mixed-methods study (SAPLAI protocol). BMJ Open. 2025 Oct 21;15(10):e105853. doi: 10.1136/bmjopen-2025-105853. PMID 41125280